CLINICAL TRIAL: NCT04388813
Title: Predictors of Severe COVID-19 Outcomes (PRESCO)
Brief Title: Predictors of Severe COVID-19 Outcomes
Acronym: PRESCO
Status: Completed | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 102293
Record Dates: First submitted 2020-05-04; First posted 2020-05-14 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a longitudinal, multi-center, observational study collecting diverse biological measurements and clinical and epidemiological data for the purpose of enabling a greater understanding of the onset of severe outcomes, primarily acute respiratory distress syndrome (ARDS) and/or mortality, in patients presenting to the hospital with suspicion or diagnosis of COVID-19. We seek to understand whether there are early signatures that predict progression to ARDS, mortality, and/or other comorbid conditions. The duration of the study participation is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative willing and able to provide informed consent
* Receiving care at a participating site
* Age 18 years old or older
* U.S. Resident
* Confirmed positive for COVID-19
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Self reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants confirmed positive for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Performance (discrimination / calibration) of models | From date of study enrollment until the date of first documented ARDS diagnosis or date of death from any cause, whichever comes first, assessed up to study end (estimated at 3 months).
  Performance (discrimination / calibration) of models that predict the risk of development of ARDS and/or mortality among COVID-19 patients who present to the hospital for evaluation and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Kim, PhD, Study Director — Verily Life Sciences LLC
Locations (8):
- United States (8):
  - The University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Inova Health Care Services, Falls Church, Virginia